CLINICAL TRIAL: NCT07115771
Title: Comparison of Ultrasound-Guided Lumbar Erector Spinae Plane Block and Adductor Canal Block on Postoperative Analgesia Management in Patients Undergoing Knee Arthroplasty
Brief Title: Comparison of Ultrasound-Guided Lumbar ESPB and ACB for Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Collaborators: Emre ULUSOY (Unknown)
Responsible Party: Principal Investigator, Mursel Ekinci, assoc prof, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bursa Şehir Hastanesi 12
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Total Knee Anthroplasty
Keywords: Postoperative Analgesia; adductor canal block; erector spinae plane block; Total Knee Anthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: he patient and the outcomes assessor who performs postoperative pain evaluation will not know the group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adductor canal block (Active Comparator): Patients will receive an adductor canal block preoperatively.
  Interventions: Other: Postoperative analgesia management
- Erector spinae plane block (Active Comparator): Patients will receive a lumbosacral erector spinae plane block in the preoperative period.
  Interventions: Other: Postoperative analgesia management

INTERVENTIONS:
Other: Postoperative analgesia management — After determining the L5-S1 level with ultrasound guidance, an 80 mm block needle (Stimuplex Ultra®, Braun, Melsungen, Germany) will be advanced in a cranio-caudal direction. Following hydrodissection, 30 ml of 0.25% bupivacaine local anesthetic solution containing 7.5 mcg of epinephrine (1:200,000) will be administered.
  Arms: Erector spinae plane block
Other: Postoperative analgesia management — After identifying the adductor canal with a high-frequency linear US probe (GE ML6-15-D Matrix Linear), 30 ml of 0.25% bupivacaine local anesthetic solution containing 7.5 mcg of epinephrine (1:200,000) will be administered into the adductor canal using an 80 mm block needle (Stimuplex Ultra®, Braun, Melsungen, Germany).
  Arms: Adductor canal block

SUMMARY:
Total knee arthroplasty (TKA) is a surgical procedure frequently associated with moderate-to-severe postoperative pain. While Adductor Canal Block (ACB) has demonstrated analgesic efficacy in TKA, the Erector Spinae Plane Block (ESPB) is also being utilized as part of multimodal analgesia for postoperative pain management in lower extremity surgeries. Currently, there is a gap in the literature as no studies have directly compared the efficacy of ACB and ESPB for pain management following TKA. The primary objective of this study is to compare the efficacy of these two analgesic methods in the context of postoperative analgesia management after total knee arthroplasty.

DETAILED DESCRIPTION:
In our clinic, various regional blocks are applied for analgesia or anesthesia purposes in many surgeries, including knee surgery. For knee surgery, adductor canal block, lumbar epidural analgesia, genicular block, erector spinae plane block, and iPACK block can be used. In our clinic, erector spinae plane block and adductor canal block are routinely applied to knee surgery patients. In our study, we aimed to contribute to the literature by comparing patient satisfaction surveys and pain follow-up in patients undergoing knee arthroplasty who received adductor canal block versus lumbosacral erector spinae plane block, both applied with PROSPECT protocols for postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent total knee arthroplasty surgery
* ASA I-II patients

Exclusion Criteria:

* Patient refusal to participate in the study
* Patients with coagulopathy
* Patients history with local anesthetic allergy or toxicity
* Patients with liver and kidney failure
* Mentally disabled patients
* Presence of infection at the injection site
* Pregnant, suspected pregnant, or breastfeeding mothers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | 0, 2, 4, 8, 16, 24 and 48 hours
  Tramadol will be prepared as 5mg/ml and patient-controlled analgesia will be administered without basal infusion, with a locking time of 20 minutes and a bolus dose of 10mg.

SECONDARY OUTCOMES:
Postoperative pain scores (Numerical rating scale) (0-meaning "no pain" to 10-meaning "worst pain imaginable") | The NRS scores of the patients will be evaluated at the postoperative 0, 2, 4, 8, 16, 24 and 48 hours.
  Postoperative 48 hours period. Patients' pain scores will be questioned at 0, 2, 4, 8, 16, 24 and 48 hours.
Global recovery scoring system (patient satisfaction scale) | The quality of recovery will be evaluated out of a total of 150 points according to the QoR-15 test to be applied at the portoperative 48th hour.
  Researchers will use the Turkish version of the Quality Improvement Survey/QoR-15. PART A: Participants will be asked by researchers how they felt in the last 24 hours.(0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent]) 1. Able to breathe easily 2. Been able to enjoy food 3. Feeling rested 4. Have had a good sleep 5. Able to look after personal toilet and hygiene unaided 6. Able to communicate with 7. Getting support from hospital doctors and nurses 8. Able to return to work or usual home activities 9. Feeling comfortable and in control 10. Having a feeling of general well-being PART B Participants will be asked by the researchers whether they have experienced any of the following in the last 24 hours. (10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor]) 11. Moderate pain 12. Severe pain 13. Nausea or vomiting 14. Feeling worried or anxious 15. Feeling sad or depressed
Determine the time to first postoperative mobilization (The Timed Up and Go - TUG test): | The Timed Up and Go (TUG) test will be performed at the 20th minute after the preoperative block.
  Place a chair in a location where walking can be observed. The area should be free of obstacles and interruptions. Measure a distance of 3 meters and draw a line on the floor at this distance. Use colored tape if available (to be clearly visible from the floor). Seat the patient in a chair, with access to their usual walking aid if applicable. Ask the patient to "start" and begin the timer. The patient stands up, walks past the 3-meter mark, turns, then walks back to the chair and sits down again. Record the time taken to complete the entire maneuver.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Tran J, Chan VWS, Peng PWH, Agur AMR. Evaluation of the proximal adductor canal block injectate spread: a cadaveric study. Reg Anesth Pain Med. 2019 Dec 25:rapm-2019-101091. doi: 10.1136/rapm-2019-101091. Online ahead of print. PMID 31879373
- [Background] Tao Y, Zheng SQ, Xu T, Wang G, Wang Y, Wu AS, Yue Y. Median effective volume of ropivacaine 0.5% for ultrasound-guided adductor canal block. J Int Med Res. 2018 Oct;46(10):4207-4213. doi: 10.1177/0300060518791685. Epub 2018 Aug 20. PMID 30124351
- [Background] Gupta A, Kaur J, Kumar R. Unilateral sacral erector spinae plane block for lower limb surgery in children. Anaesth Rep. 2022 Dec 14;10(2):e12199. doi: 10.1002/anr3.12199. eCollection 2022 Jul-Dec. PMID 36530341
- [Background] Browne W, Nair BKR. The Timed Up and Go test. Med J Aust. 2019 Jan;210(1):13-14.e1. doi: 10.5694/mja2.12045. Epub 2018 Dec 28. No abstract available. PMID 30636313
- [Background] Diwan S, Nair A. Lumbar erector spinae plane block obtunding knee and ankle reflexes. Saudi J Anaesth. 2021 Apr-Jun;15(2):222-224. doi: 10.4103/sja.SJA_79_20. Epub 2021 Apr 1. PMID 34188648
- [Background] Kaya C, Dost B, Tulgar S. Sacral Erector Spinae Plane Block Provides Surgical Anesthesia in Ambulatory Anorectal Surgery: Two Case Reports. Cureus. 2021 Jan 9;13(1):e12598. doi: 10.7759/cureus.12598. PMID 33585088
- [Background] Selvi O, Azizoglu M, Temel G, Tulgar S, Chitneni A, Cinar EN, Ozer Z, Gurkan Y. Translation and Validation of the Turkish Version of the Quality of Postoperative Recovery Score QoR-15: A Multi-Centred Cohort Study. Turk J Anaesthesiol Reanim. 2022 Dec;50(6):443-448. doi: 10.5152/TJAR.2022.21417. PMID 36511494